CLINICAL TRIAL: NCT01200576
Title: A Prospective Observational Study of the Clinical Performance of Zarin in Madagascar
Status: Completed | Type: Observational
Sponsor: FHI 360 (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Marie Stopes International (Other)
Responsible Party: Sponsor
Other Study IDs: 10225
Record Dates: First submitted 2010-09-10; First posted 2010-09-13 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Long-term and Permanent Contraceptive Methods
Keywords: CRF: Case Report Form; DM: Data Management; FHI: FHI (formerly known as Family Health International); IRB: Institutional Review Board; IUD: Intra-uterine Device; LTPM: Long-term and Permanent Contraceptive Methods; MSI: Marie Stopes International; MSM: Marie Stopes Madagascar; PHSC: Protection of Human Subjects Committee; PI: Principal Investigator; SAE: Serious Adverse Event; Sino-Implant (II); SOP: Standard Operating Procedure; Zarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: healthy volunteers

SUMMARY:
This one-year observational study will monitor the contraceptive effectiveness, safety and acceptability of Zarin during the first year of use after the method has been approved for public use in Madagascar. It will be implemented by Marie Stopes Madagascar with technical support from Marie Stopes International and FHI. 300 women of reproductive age who selected Zarin as their primary method of contraception will be enrolled in the study at the MSM outreach sites and static clinics.

DETAILED DESCRIPTION:
This one-year observational study will monitor the contraceptive effectiveness, safety and acceptability of Zarin during the first year of use after the method has been approved for public use in Madagascar. It will be implemented by Marie Stopes Madagascar with technical support from Marie Stopes International and FHI. 300 women of reproductive age who selected Zarin as their primary method of contraception will be enrolled in the study at the MSM outreach sites and static clinics.

ELIGIBILITY:
Inclusion Criteria:

* be a participant of the MSM service evaluation and continue using Zarin at 3 months
* agree at the time of Zarin insertion to be contacted regarding an opportunity to participate in more research related to the implant

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: healthy women of any age
Sampling Method: Probability Sample
Enrollment: 621 (Actual)
Dates: Start 2010-10; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The cumulative probability of pregnancy through one year | 1 year
Prevalence and incidence rate of adverse events | 1 year
Prevalence and incidence rates of immediate and delayed complications associated with insertion or removal | 1 year
The cumulative probability of early discontinuation through one year | 1 year
Reasons for discontinuation | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Odile Hanitriniaina, MD, Principal Investigator — Marie Stopes International; Kristen Hopkins, Study Chair — Marie Stopes International; Tania Boler, Principal Investigator — Marie Stopes International; Markus Steiner, Ph.D., Principal Investigator — FHI 360
Locations (1):
- Marie Stopes Madagascar Mobile Outreach Sites and Static Clinics, Madagascar, Madagascar